CLINICAL TRIAL: NCT03591237
Title: Mindfulness-based Cognitive Therapy for Pain in Cancer Patients After Primary Treatment: An Open Implementation Trial
Brief Title: MBCT for Cancer Patients in Follow-Up
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MBCT-late effects 2018
Record Dates: First submitted 2018-03-26; First posted 2018-07-19 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Pain Management
Keywords: cancer; late effects; pain
MeSH Terms: conditions — Agnosia; Neoplasms; Pain | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MBCT (Experimental): As patients with significant pain are identified and accept the offer of receiving 'Mindfulness-Based Cognitive Therapy' (MBCT) for pain, they will be consecutively included in groups of 12-20 participants. The patients will participate in eight weekly two hour group sessions and will be asked to do an additional 45 minutes of daily training at home.
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy — The patients participate in eight weekly group sessions of two hours each and will be asked to do an additional 45 minutes of daily training at home. The participants will be asked to record their home training to allow assessment of their adherence to the intervention. Generally, the program corresponds to the manualized MBCT program, but with adaptations that take into account the special needs of cancer patients, including shorter sessions, shorter yoga exercises and the omission of the all-day session. The sessions include psychoeducation and formalized mindfulness exercises with focus on the participants' here-and-now experience of their pain.

SUMMARY:
The objectives of the present study are: 1) to executing the practical implementation in an oncology department of MBCT for patients who have completed their primary treatment and experience significant cancer- and cancer-treatment-related pain, 2) to evaluate effects on pain and well-being, 3) to explore patient satisfaction with the intervention offered, and 4) to explore possible organizational and individual physical, mental and socio-economic barriers for implementation in relation to drop-outs.

DETAILED DESCRIPTION:
International research shows that untreated or under treated pain among cancer patients after completion of therapy is a common problem with substantial negative impact on the patients' quality of life and mental and physical function.These challenges have increased interest in psychological pain therapy and among the available methods of psychological intervention, mindfulness-based interventions (MBI) are of particular interest. MBI appears to be particularly relevant for pain, as mindfulness focuses, through different meditation exercises, on concentrating attention on here-and-now experiences and supporting new ways of addressing physical sensations and emotional discomfort, characterized by greater acceptance and openness. MBI has been shown effective in treatment of nonmalignant chronic pain. . Patients seen by all four diagnosis teams at the Oncology Department at AUH are screened for pain (0-10 NRS) in connection with their final consultation with the oncologist. Patients with a pain score of ≥ 4 on one or more of the four pain dimensions questions receive a folder describing MBCT and the treatment plan and are encouraged to contact the MBCT team for more information and scheduling of an interview. If the patient, after initial information either by phone or after the first interview decline the offer to participate, but are willing to be contacted for the purpose of gathering more information about their reasons for not participating, we will send them a brief questionnaire concerning their pain and their reasons for choosing to decline the offer, to complete online. They are also asked to give their permission to collect the same information after three months. All data are collected and registered with REDCap, a high data security project administration system administered by Aarhus University's Clinical Trial Unit. The patients will participate in eight weekly two hour group sessions and will be asked to do an additional 45 minutes of daily training at home. The participants will be asked to record their home training to allow assessment of their adherence to the intervention. The program corresponds to the manualized MBCT program, but with adaptations that take into account the special needs of cancer patients, including somewhat shorter sessions, shorter yoga exercises, and the omission of the all-day session. The sessions include psychoeducation and formalized mindfulness exercises with focus on the participants' here-and-now experience of their pain. The aim of the present project is to evaluate the practical implementation of MBCT, with focus on: 1) the observed effects on pain (primary outcome parameter), 2) effects on quality-of-life (QoL) and on other cancer and cancer-treatment-related late effects associated with pain (secondary outcome parameter), 3) possible barriers for continued participation in the program (drop-out), 4) patient experience and satisfaction with the intervention and its organizational/practical implementation, 5) staff's experience of screening procedure and implementation, and 6) collection of data for use in the evaluation of effects, costs, and savings. For use in the evaluation, the patients complete questionnaires prior to the first session (T1), immediately after the last session (T2), and at a six-month follow-up (T3).

ELIGIBILITY:
Inclusion Criteria:

* >18 yrs. of age
* completed primary cancer treatment
* experiencing moderate to severe pain >4 (11-point NRS)

Exclusion Criteria:

* incomplete chemotherapy or radiation therapy
* serious psychiatric diagnoses eg. psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity assessed by NRS | Change in pain intensity from baseline (day 0) to post-intervention (up to 30 weeks after baseline)
  Pain intensity during the last week is assessed by a 11-point numeric rating scale (NRS), range 0-10. (0=no pain, 10= worst pain ever).
Pain interference assessed by NRS | Change in pain interference from baseline (day 0) to post-intervention (up to 30 weeks after baseline)
  Pain interference with daily activities during the last week is assessed by a 11-point numeric rating scale (NRS), range 0-10. (0=no interference, 10=maximal interference).

SECONDARY OUTCOMES:
Pain quality assessed by the McGill Pain Questionnaire (SF-MPQ-2) | Change in pain quality from baseline (day 0) to post-intervention (up to 30 weeks after baseline)
  Pain quality is assessed by the McGill Pain Questionnaire, which consists of 22 items representing different descriptors of pain. Each item is rated based on a 0-10 scale (0=no pain, 10=worst pain ever) during the last week. The questionnaire comprises of four parts, including continuous, intermittent, neuropathic and affective pain.
Pain burden assessed by NRS | Change in pain burden from baseline (day 0) to post-intervention (up to 30 weeks after baseline)
  Pain burden is assessed by a 11-point numeric rating scale (NRS), range 0-10 "How burdensome have your pain been during the last week" (0=not burdensome, 10=very burdensome).
Cancer-related quality of life assessed by EORTC-QLQ-C30 | Change in cancer-related quality of life from baseline (day 0) to post-intervention (up to 30 weeks after baseline)
  Cancer-related quality of life is assessed with the European Organisation for Research and Treatment of Cancer's quality of life questionnaire (EORTC-QLQ-C30), which consists of 30 items.
Health-related quality of life assessed by the EQ-5D-3L | Change in health-related quality of life from baseline (day 0) to post-intervention (up to 30 weeks after baseline)
  Health-realted quality of life is assessed by the EQ-5D, which consists of 5 items, measuring five dimensions of health status: mobility, self-case, usual activities, apin/discomfort, anxiety/depression. Each item is rated by marking a statement representing values at three levels 1-3. Higher scores indicate lower levels of quality of life.
Well-being assessed by the WHO-5 | Change in well-being from baseline (day 0) to post-intervention (up to 30 weeks after baseline)
  Well-being is assessed by the World Health Organization Well-Being Index (WHO-5), which consists of 5 items. Each item is rated on a 6-point Likert scale, ranging from 0-5. Higher scores indicate higher levels of well-being.
Fear of cancer recurrence assessed by the FCRI-SF | Change in fear of cancer recurrence from baseline (day 0) to post-intervention (up to 30 weeks after baseline)
  Fear of cancer recurrence is assessed with the Fear of Cancer Recurrence Inventory - Short Form (FCRI-SF), which consists of 9 items. Each item is rated on a 5-point Likert scale, ranging from 0-4. Higher scores indicate higher levels of fear of cancer recurrence.
Symptoms of depression assessed by the BDI | Change in depression symptoms from baseline (day 0) to post-intervention (up to 30 weeks after baseline)
  Depressive symptoms are assessed by the Beck Depression Index (BDI), which consists of 21 items. Each item is rated by marking a statement representing values from 0-3. Higher scores indicate higher levels of depression symptoms.
Sleep quality assessed by the ISI | Change in sleep quality from baseline (day 0) to post-intervention (up to 30 weeks after baseline)
  Sleep difficulties are assessed by the Insomnia Severity Index (ISI), which consists of 7 items. Each item is rated on a 5-point Likert scale, ranging from 0-4. Higher scores indicate higher severity of insomnia.

OTHER OUTCOMES:
Pain catastrophizing assessed by the PCS | Session-by-session change in pain catastrophizing from baseline (day 0) to post-intervention (up to 30 weeks after baseline)
  Pain catastrophizing is assessed by the Pain Catastrophizing Scale (PCS), which consists of 13 items. Each item is rated on a 5-point Likert scale (0=not at all, 4=all the time). Higher scores indicate higher levels of pain catastrophizing.
Experiential avoidance assessed by the BEAQ | Session-by-sessions change in experiential avoidance from baseline (day 0) to post-intervention (up to 30 weeks after baseline)
  Experiential avoidance is assessed by the Brief Experiential Avoidance Questionnaire (BEAQ), which consists of 15 items. Each item is rated on a 6-point Likert scale, ranging from 1=strongly disagreee to 6=strongly agree. Higher scores indicate higher levels of experiential avoidance.
Mindfulness assessed by the FFMQ | Session-by-session change in mindfulness from baseline (day 0) to post-intervention (up to 30 weeks after baseline)
  Mindfulness is assessed by the Five Facet Mindfulness Questionnaire (FFMQ), which consists of 39 items. The questionnaire measures five mindfulness facets: acting with awareness, describing, nonjudging of inner experience, nonreactivity to inner experience, observing. Each item is rated on a 5-point Likert scale (1=never or rarely true, 5=very often or always true). Higher scores indicate higher levels of mindfulness.
Self-compassion assessed by the SCS | Session-by-session change in self-compassion from baseline (day 0) to post-intervention (up to 30 weeks after baseline)
  Self-compassion is assessed by The Self-Compassion Scale - Short form (SCS-SF), which consists of 12 items. Each item is rated on a 5-point Likert scale (1=almost never, 5=almost always). Higher scores indicate higher levels of self-compassion.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zachariae, DMSCi, Principal Investigator — University of Aarhus
Locations (2):
- Denmark (2):
  - Aarhus University, Aarhus, Jylland
  - Dept of Oncology, Aarhus University Hospital, Aarhus, Jylland

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-02): https://cdn.clinicaltrials.gov/large-docs/37/NCT03591237/Prot_SAP_000.pdf